CLINICAL TRIAL: NCT03219671
Title: A Phase 2 Study of Nivolumab Plus Ipilimumab in Previously Treated Classical Kaposi Sarcoma (CKS)
Brief Title: Nivolumab and Ipilimumab in Classical Kaposi Sarcoma (CKS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alona Zer (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Alona Zer, Senior Physician, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-937; 0095-17-RMC (Other: Rabin Medical Center)
Record Dates: First submitted 2017-06-26; First posted 2017-07-17 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Classic Kaposi Sarcoma
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- nivolumab plus ipilimumab (Experimental): nivolumab 240mg every 2 weeks plus ipilimumab 1 mg/kg every 6 weeks
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — nivolumab 240mg every 2 weeks
Drug: Ipilimumab — ipilimumab 1 mg/kg every 6 weeks

SUMMARY:
A Phase 2 study of nivolumab plus ipilimumab in previously treated classical Kaposi Sarcoma (CKS)

DETAILED DESCRIPTION:
A prospective, single arm, interventional study. All patients will receive IV nivolumab 3mg/kg every two weeks and ipilimumab 1mg/kg every 6 weeks. Patients will be treated until disease progression or intolerable toxicity for a maximal period of two years, with an option to re-initiate therapy upon progression in patients with prior documented response to investigational therapy (unless treatment was held for progression of disease).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed KS
* Age > 18
* ECOG PS < 2
* At least one prior treatment modality (palliative radiation or chemotherapy)
* Measurable disease as defined by RECIST version 1.1 by physical exam and/or PET-CT (previously irradiated lesions should not be counted as target lesions).

Exclusion Criteria:

* Patients with HIV-related KS or HIV positive serology.
* Ongoing immunosuppressive therapy
* Active autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 6-months
  overall response rate (ORR)

SECONDARY OUTCOMES:
PFS rate | 6-months
  6-months PFS rate
Safety - Incidence of Treatment-Emergent Adverse Events according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, Version 4.0 (CTCAE v4) | during the study, through study completion, an average of 1 year
  Patients will be evaluated for treatment related adverse events (AEs) on each visit during study participation and toxicity will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, Version 4.0 (CTCAE v4).
Tolerability - treatment related adverse events (AEs) that caused study drug interruption and discontinuation | during the study, through study completion, an average of 1 year
  Patients will be evaluated for treatment related adverse events (AEs) that caused study drug interrupption and discontinuation.

OTHER OUTCOMES:
Exploratory Biomarkers | 6-months
  including, but not limited to proteins and/or genes involved in regulating immune responses (eg PD-L1, IDO1, KYN and MSI status).

CONTACTS AND LOCATIONS:
Overall Officials: Alona Zer, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No